CLINICAL TRIAL: NCT02911272
Title: Labour Outcomes With Partograph Action Line Placement at 2 Hour Versus 4 Hours: A Randomised Controlled Trail
Brief Title: Best Partograph Action Line to Prevent Prolonged Labour
Acronym: Partograph
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Benin (Other)
Responsible Party: Principal Investigator, Augustine A.E Orhue, Principal investigator, University of Benin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UBenin
Record Dates: First submitted 2016-09-14; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Prolonged First Stage Labor - Prevention
Keywords: Partograph; Best action line; Prolonged labour prevention
MeSH Terms: interventions — Oxytocin; Amniotomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2-hour group (Active Comparator): Augmentation of labour at 2-hour action line on the labour partograph
  Interventions: Device: 2-hour action line on WHO modified partograph; Drug: Oxytocin; Procedure: Forewater amniotomy
- 4-hour group (Experimental): Augmentation of labour at 4-hour action line on the labour partograph
  Interventions: Drug: Oxytocin; Procedure: Forewater amniotomy; Device: 4-hour action line on WHO modified partograph

INTERVENTIONS:
Device: 2-hour action line on WHO modified partograph — observations and findings in a woman in labour are recorded on this device (WHO modified partograph) in a graphic format in which the action line is located 2-hour from the alert line
  Arms: 2-hour group
Drug: Oxytocin — Oxytocin augmentation of slow labour progress at the respective action line location on the WHO modified partograph
Procedure: Forewater amniotomy — Forewater amniotomy at the vaginal examination confirming active phase labour
  Other Names: Artificial rupture of membrane
Device: 4-hour action line on WHO modified partograph — observations and findings in a woman in labour are recorded on this device (WHO modified partograph) in a graphic format in which the action line is located 4-hour from the alert line
  Arms: 4-hour group

SUMMARY:
Objective: To compare active labour outcomes in nulliparous women at term supervised with a partograph with the action line placed at either 2 hours or 4 hours and to determine whether the 2-hour action line placement is better for the prevention of prolonged labour.

Design: Randomised controlled trial.

Setting: A university teaching hospital in Nigeria.

Population: Nulliparous women in labour at term.

Method: Nulliparous women in labour were randomly supervised with a partograph with the action line placed at 2 hours (n=320) or 4 hours (n=320). Oxytocin augmentation, when required, was used only at the 2-hour (n=87) or 4-hour (n=61) action lines. Progress monitoring was the same in both groups.

Main outcome measure: The primary outcome measure was the prolonged labour rate. The secondary outcome measures were the mode of delivery and neonatal outcome.

DETAILED DESCRIPTION:
Materials and methods

This prospective, randomised controlled study was conducted from April 2008 to April 2013. The labour ward staff had very good knowledge of how to use the partograph, and partographs were routinely supplied in the labour ward. The department had a management protocol for the use of the partograph for labour supervision of all parturients in labour. In addition, an audited review of how labour was managed in all parturients occurred every morning on all workdays to assess compliance with the management protocol, which ensured the continuous instruction of all staff in partograph use for labour supervision.

At the time of admission, the study participants were nulliparous, between 37 and 42 weeks gestation, in the spontaneous active phase of labour with intact fetal membranes and had singleton, cephalic-presenting fetuses. The exclusion criteria were prior antepartum haemorrhage, medical disorders in pregnancy and poor fetal growth in pregnancy. All the women who fulfilled the inclusion criteria during the antenatal period at approximately 34-36 weeks were selected, participated in an informative discussion about the study and signed a written consent. The study was approved by the UBTH research and ethics committee after a review of the study protocol and informed consent details. However, final inclusion in the study was limited to previously selected women who arrived at the labour ward at term in spontaneous active-phase labour with intact fetal membranes and still had no exclusion criteria. Upon presenting at the labour ward and being confirmed to be in active labour, the consenting women were randomised to either of two study arms: labour supervision with composite partograph action line location at 2 hours or 4 hours from the alert line by the physician but blinded to the participants. Allocation to the study arms was performed using consecutively numbered, sealed, opaque envelopes with a randomised sequence using a computer random number generator by a statistician not involved with care. A sample size determination for a 2-hour versus a 4-hour oxytocin augmentation of labour with a type 1 error (alpha) of 10% and a type II error (beta) of 20% together with a power of 80% and a level of significance of 0.05 was performed on the basis of a previous study on the effects of different partograph action lines on birth outcomes. Recruitment into each arm of the study was calculated to require 320 participants. The enrolment of women in the study was continued until a sample size of 320 was achieved in each study group, the 2-hour or 4-hour action line. There were therefore no exclusions.

Data and statistical analysis

Collected data were checked for completeness and analysed using SPSS version 17 (SPSS Inc., 233 South Wackor Drive, Chicago, Illinois 60606-6412, USA). Bivariate analyses were performed using a chi-square test for differences in proportion between the 2-hour and 4-hour lines for categorical variables, and odds ratios (ORs) and the respective confidence intervals were calculated. Continuous variables were compared using unpaired t-tests. A p-value of <0.05 was considered indicative of statistical significance.

According to the departmental protocol for spontaneous labour management, active-phase labour was defined as at least one progressive contraction at every 10-minute interval in a parturient at term with cervical os confirmed as 4cm or above. The fetal membranes were instantly ruptured at the same vaginal examination (VE), which confirmed active-phase labour in all parturients to facilitate cervical os dilatation at 1 cm per hour because intact fetal membranes cause slow labour progress during active-phase labour. Findings from admission or first VE during active labour and other feto-maternal vital signs were recorded on the partograph. The feto-maternal vital signs were subsequently recorded hourly on the partograph.

The timing of the repeat VE depended on the location of the action line on the partograph, to which the parturient was randomly allocated. For the women allocated to the 2-hour action line partograph, repeat VEs occurred every 2 hours. Women in the 4-hour group received repeat VEs every 4 hours unless the cervical os dilatation at the first VE was 7cm or above, in which case the repeat VE was performed earlier than 4 hours. The cervical os dilatations from the first and all subsequent VE findings were plotted on the partograph to show the graph of cervical os dilatation. When the cervical os dilatation progress did not cross the alert line, the progress was regarded as normal, and the subsequent care and delivery was performed by the midwife or junior obstetrics staff resident doctor. When the cervical os dilatation progress plotted on the partograph crossed the alert line, the midwife transferred the case to the obstetric team for subsequent care until delivery.

Although all the parturients were admitted to the labour ward and had their first VE conducted by a midwife and recorded on the partograph, no midwife or obstetric resident staff of a status below a senior obstetric resident was allowed to perform a VE more than twice within 2 to 4 hours on any parturient in active-phase labour. The need for a third VE by the midwife or junior obstetric staff (other than a senior resident) was considered an indication to transfer the parturient to the care of more senior obstetric staff with the skill to manage long-duration active-phase labour. This strategy ensured the involvement of the senior obstetric staff in the treatment of women who remained in active-phase labour. Oxytocin augmentation as a treatment for slow labour progress was instituted only when the 2-hour or 4-hour action line was crossed, not by the quality or frequency of uterine contractions as assessed by any method. The oxytocin base mixture and titration regimen in this study was as by the departmental protocol.

A parturient on oxytocin labour augmentation was assigned a midwife to act as companion and to monitor the infusion regimen. The maximum duration of oxytocin augmentation was 8hours in the absence of fetal distress. When augmentation had occurred for over 4 hours, the senior obstetric resident managing the case was required to inform the consultant on call duty, who was also required to be involved in all caesarean delivery-related decisions for any parturient in labour, especially if there had been augmentation of labour. According to this protocol, the partograph in our setting was used as a tool for the deployment of the labour ward staff for the management of active-phase labour in cooperation between the midwives and obstetric staff. By this arrangement, parturients whose labour progress did not cross the alert line were managed and delivered by the midwives, while the parturients whose labour progress crossed the action line were passed to the care of the more senior and experienced obstetric staff for effective and efficient labour care. Prolonged labour, as defined by the departmental protocol and in this study, was defined as an active-phase labour duration of over 12 hours.

The third stage of labour was actively managed to minimise blood loss. On the first day post-delivery, women who had vaginal delivery were interviewed using the likert scale score model regarding their satisfaction with the intervention based on the partograph action line placement and analysis was by one of the authors who was blinded to the action line placement. Those who delivered by c/s had their interview conducted on the third day post-delivery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy nulliparous patients at term in spontaneous active phase labour with singleton pregnancies and intact fetal membranes at first vaginal examination in labour ward

Exclusion Criteria:

* Multiparous patients
* Multiple pregnancies
* Pre-existing medical conditions complicating pregnancy
* Non-cephalic presenting fetus at term
* Prelabour rupture of membrane at term
* Preterm labour
* Poor fetal growth in pregnancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2008-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Duration of active phase labour | At the point of each patient's delivery within 24 hours from onset of labour
  Time spent from admission in active phase labour till point of delivery expressed in hours

SECONDARY OUTCOMES:
Mode of delivery | within 24 hours from onset of labour
  Vaginal delivery or cesarean section
Neonatal Asphyxia | at the point of delivery within 24 hours from onset of labour
  Apgar score of the neonates of less than 7 assessed at the first minute of life

CONTACTS AND LOCATIONS:
Overall Officials: Augustine AE Orhue, FRCOG, Principal Investigator — University of Benin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orhue A, Oseihie II, Aziken M, Ande B. Randomized controlled trial of labor outcomes with action line placement at 2 hours versus 4 hours on the partograph. Int J Gynaecol Obstet. 2020 Jul;150(1):64-71. doi: 10.1002/ijgo.13144. Epub 2020 Apr 17. PMID 32301113